CLINICAL TRIAL: NCT01692808
Title: Bioavailability of Vitamin D in Children and Adolescents With Crohn's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jantchou Prevost, Professor, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP2012042
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Crohn's Disease
Keywords: Crohn; vitamin D; remission; inflammation; tolerance
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Exclusive Enteral Nutrition (No Intervention): This group is one of the non interventional group. As enteral nutrition is one of the usual therapy of Crohn disease at diagnosis.
- EEN + Vitamin D3 3000 UI daily (Experimental): Exclusive Enteral Nutrition + Vitamin D3 3000 UI daily for one month This arm will be one of the two experimental arms.
  Interventions: Drug: Vitamin D3 3000 UI daily
- Corticosteroïd (No Intervention): Corticosteroids (1mg/kg/day) associated with usual vitamin and calcium supplementation: vitamin D 800 IU of vitamin D3 + 1000 mg calcium per day) for one month
- Corticosteroids + Vitamin D3 4000 UI (Experimental): Corticosteroids (1mg/kg/day) associated with vitamin D3 4000 UI daily and calcium 1000 mg daily for one month
  Interventions: Drug: Vitamin D3 4000 UI daily
- Vitamin D3 4000 UI (Experimental): Vitamin D3 4000 UI /day . This arm is intended for those children in remission with or without immunosuppressant. Vitamin D will be administered in adjunction to usual therapy.
  Interventions: Drug: Vitamin D3 4000 UI daily

INTERVENTIONS:
Drug: Vitamin D3 3000 UI daily — Vitamin D3 will be administered as an adjunct to corticosteroids or enteral nutrition at the doses of 3000 UI daily or 4000 UI daily
  Other Names: Cholecalciferol
  Arms: EEN + Vitamin D3 3000 UI daily
Drug: Vitamin D3 4000 UI daily — This arm is intended for those at diagnosis treated with Corticosteroid or in Remission
  Other Names: Cholecalciferol
  Arms: Corticosteroids + Vitamin D3 4000 UI; Vitamin D3 4000 UI

SUMMARY:
The purpose of this study is to determine if high doses of vitamin D3 administered orally as adjunct therapy to children with Crohn's disease could improve the outcome of the disease.

DETAILED DESCRIPTION:
Background : Crohn's disease is a chronic inflammatory condition affecting all segments of the digestive tract from the mouth to the anus. This condition is associated with an increased risk of relapses throughout the course of the disease. Nearly 25% of patients with Crohn's disease are in the pediatric age range. Many epidemiological data are in favor of an increase incidence of pediatric Crohn's disease. Environmental factors could explain this increased incidence. Among them sunlight exposure and vitamin D deficiency have been suggested by many authors.

Vitamin D, in addition to its action on bone metabolism, exerts an anti-inflammatory effect by modulating the innate and acquired immune system. The biological effect of high doses of vitamin D administered orally have not been extensively studied in children with Crohn's disease. In these patients, the absorption and bioavailability of vitamin D may be altered in relation with mucosal lesions.

Objective :

Thus our aim is to investigate the effect of high doses of vitamin D3 administered orally as an adjunct therapy to children with newly diagnosed pediatric Crohn diseases or children in remission.

Methods : In this Prospective study 40 children will be enrolled and followed up for a duration of one month. The administration of vitamin D 3000 IU or 4000 IU per day will be considered as an adjunct to conventional therapy (steroids or enteral nutrition for patients at diagnosis or immunosuppressants for patients in remission).

Analysis:

1. Tolerance will be assessed during weekly visits by a brief questionnaire and blood tests.
2. Efficacy will be assessed by monitoring the change in fecal and blood inflammatory markers.
3. Change in the immunological status will be assessed by measuring the following parameters :

   * T lymphocyte count CD3, CD4, CD8, and invariant Natural Killer T cell, Treg.
   * Proliferation and activation of CD4 and CD8 T lymphocytes induced by anti-CD3 antibody activator (OKT3). The activation will be evaluated by dosing CD25 and the proliferation by the study of cell cycle after 3 days of culture of total blood culture.
   * The culture supernatants will be collected and frozen for subsequent analysis of cytokines Th1 and Th2 (IFN, IL2, IL4, IL13) with Affymetrix method that allows simultaneous determination of multiples cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Age between 10 and 18 years
* Crohn's disease diagnosed by usual clinical and endoscopic criteria
* Recent (less than one week) blood test with results of : Albumin, sedimentation rate, hematocrit

Exclusion Criteria:

* Known renal or cardiac malformation
* Disorders of phospho-calcic metabolism and vitamin D
* Intake of vitamin D supplementation in the last three months prior to enrollment
* Current intake of medications known to interfere with the metabolism of calcium, phosphate and vitamin D *

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events after one month | up to 1 month
  Tolerance will be assessed weekly by measuring clinical adverse events in relation with high blood level of 25 hydroxy vitamin D.
  Biological measures will also be performed including : Circulating level of Calcium, phosphorus, PTH.

SECONDARY OUTCOMES:
Decrease of inflammatory parameters | Baseline and 1 month
  Evaluate the change from baseline in effect in blood and fecal inflammatory parameters (erythrocyte sedimentation rate, C-reactive protein, faecal Calprotectin).
Immunological changes | Baseline and 1 month
  Evaluate the change from baseline in immunological parameters (lymphocytes CD3, CD4, CD8, Treg and iNKT, proliferation and activation of CD4 and CD8).
Bioavailability | Baseline, after 24 h and then weekly for one month
  The bioavailability will be assessed by measuring the level of 25 hydroxy vitamin D at baseline then 24 hours after the first administration of vitamin D then weekly up to one month and compare this level to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Prevost Jantchou, MD, PHD, Principal Investigator — mother-child university hospital Ste. Justine Montreal-Canada
Locations (1):
- Mother-child university hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Jantchou P, Clavel-Chapelon F, Racine A, Kvaskoff M, Carbonnel F, Boutron-Ruault MC. High residential sun exposure is associated with a low risk of incident Crohn's disease in the prospective E3N cohort. Inflamm Bowel Dis. 2014 Jan;20(1):75-81. doi: 10.1097/01.MIB.0000436275.12131.4f. PMID 24247650
- [Result] Nerich V, Jantchou P, Boutron-Ruault MC, Monnet E, Weill A, Vanbockstael V, Auleley GR, Balaire C, Dubost P, Rican S, Allemand H, Carbonnel F. Low exposure to sunlight is a risk factor for Crohn's disease. Aliment Pharmacol Ther. 2011 Apr;33(8):940-5. doi: 10.1111/j.1365-2036.2011.04601.x. Epub 2011 Feb 20. PMID 21332762